CLINICAL TRIAL: NCT03450148
Title: Acceptability and Feasibility of Self Administered Aversive Therapy for Smoking Cessation
Brief Title: Aversive Therapy for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nipam Shah, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F23234543
Record Dates: First submitted 2018-02-13; First posted 2018-03-01 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2020-09

CONDITIONS: Smoking Cessation
Keywords: aversive therapy
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pavlok wristband with electric stimulus (Experimental): Participants in intervention group will wear wristband and will get a slight electric stimulus when they press the device
  Interventions: Other: Pavlok wristband with electric stimulus
- Pavlok wristband without electric stimulus (Placebo Comparator): Participants in control group will wear wristband and will not get a slight electric stimulus when they press the device
  Interventions: Other: Pavlok wristband without electric stimulus

INTERVENTIONS:
Other: Pavlok wristband with electric stimulus — it is a device for various behavior modifications in the form of wristband which participants will wear on the wrist. Device has maximum voltage of 0-500 volts, delivers a electric stimulus for a maximum of 1 sec and average duration of 0.2 secs
  Arms: Pavlok wristband with electric stimulus
Other: Pavlok wristband without electric stimulus — it is a device for various behavior modifications in the form of wristband which participants will wear on the wrist. Participants will not receive any electric stimulus since this feature will be turned off.
  Arms: Pavlok wristband without electric stimulus

SUMMARY:
The purpose of this research study is to test a new way to help people quit smoking. The PI will test acceptability and feasibility of a new device called Pavlok wearable wrist band. Participants will be smokers who are highly motivated to quit. Participants will be randomized into intervention and control groups.

DETAILED DESCRIPTION:
The participants will be evaluated after 1 week and assessed for their ongoing participation and commitment to the study. Those still interested and eligible will be randomized to two groups described below and will continue the study for 3 more weeks. There will be follow up surveys at various time points while wearing the wristband (1 week, 2 week, 3 weeks) and a final survey at T=3 months.

The intervention group will continue to wear the wristband and the wristband will deliver a slight electric stimulus every time it is pressed.

The placebo group will wear continue to press the button on the wristband but it will not give a slight electric stimulus when pressed. Both groups will wear the device for a total of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker (defined by the Center for Disease Control as an "adult who has smoked 100 cigarettes in his or her lifetime and who currently smokes cigarettes ". This will be determined based on participant baseline survey.
* Interested in quitting (contemplation stage and beyond, as defined by serious consideration of quitting smoking in the next 30 days
* Subject is equal to or greater than 19 years old
* Considers themselves "tech savvy" (based on self reported 5 point likert scale)
* Must have a smart phone with blue tooth capabilities
* Willing to receive aversive therapy if assigned to this group.

Exclusion Criteria:

* Anyone with a diagnosed arrhythmia or with a pacemaker or with a phobia or history of psychosis.
* Non-English speaking caregivers
* Lives outside of contiguous United States

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Participants acceptability: short customized survey | T=0 to 3 months
  Participants' acceptability/satisfaction will be assessed using a short customized survey. The survey will include 8 questions with options ranging from strongly agree to strongly disagree for five questions and ranging from satisfaction to dissatisfaction for the remainder 3 questions. Each question will be evaluated individually.
Evaluate the dropout among participants | T=0 to 3 months
  Number of participants dropped out from time of randomization. Dropout is defined as missing two follow up assessments.
Enrollment percentage of eligible participants | Baseline to T=0
  PI will evaluate the percentage of participants that were enrolled after the 1 week run in period.
Percentage of time wristband worn by participants | T=0 to one week
  PI will evaluate the percentage of time the wristband is worn. Instructions will be given to wear the wristband all of the waking hours.
Percentage of time wristband worn by participants | from one week to two weeks
  PI will evaluate the percentage of time the wristband is worn. Instructions will be given to wear the wristband all of the waking hours.
Percentage of time wristband worn by participants | from two week to three weeks
  PI will evaluate the percentage of time the wristband is worn. Instructions will be given to wear the wristband all of the waking hours.
Participants satisfaction: short customized survey | T=0 to 3 months
  Participants' acceptability/satisfaction will be assessed using a short customized survey. The survey will be a Likert scale and will include 2 questions with options ranging from satisfied to dissatisfied (with 1 indicating satisfaction and 5 indicating dissatisfaction). One other question is a likert scale with options ranging from 1-3 with 1 indicating the device was very useful and 3 indicating the device was not at all useful. A higher score indicates a worse outcome (less satisfaction with the device). Each question will be evaluated individually.

SECONDARY OUTCOMES:
Percentage of participants that made a quit attempt | From T=0 to one week
  PI will evaluate the percentage of participants that made a quit attempt as defined by absence of smoking for more than 24 hours in the previous seven days. This will be assessed through the follow up survey given at various intervals.
Percentage of participants that made a quit attempt | From T=1 week to 2 weeks
  PI will evaluate the percentage of participants that made a quit attempt as defined by absence of smoking for more than 24 hours in the previous seven days. This will be assessed through the follow up survey given at various intervals.
Percentage of participants that made a quit attempt | From T= 2 weeks to 3 weeks
  PI will evaluate the percentage of participants that made a quit attempt as defined by absence of smoking for more than 24 hours in the previous seven days. This will be assessed through the follow up survey given at various intervals.
Average Degree of smoking reduction | From baseline to 3 months
  PI will evaluate the average percentage of smoking reduction. This will be quantified by the average number of cigarettes smoked at baseline compared to the average number of cigarettes smoked at 3 months. This will be assessed via the "Follow survey".
Percentage of participants who had cessation of smoking. | T=0 to T= 3 weeks
  P will evaluate the percentage of participants who had cessation of smoking, as defined by the absence of smoking in the previous 30 days. This will be evaluated by the "Three month Questionnaire"
Before and after smoking self-efficacy score | Baseline to 3 months
  The PI will evaluate the self-efficacy of the participant as evaluated by the "Baseline Smoking self-efficacy scale Short form". There are 9 questions which will assess the confidence of the participant to not smoke.The investigators will use Likert scale for each question which assesses the participants confidence to "not smoke" in various circumstances. The answers range from 1 to 5 with 1 indicating "not at all confident" and 5 indicating "extremely confident". The overall score for each participant will be calculated by sum of scores from all items. This score for individual subscales will be calculated by sum item scores so that the total score will range from 9 to 45, with a lower score indicating a worse outcome i.e. less confidence to not smoke).
Stage of change | From baseline until 3 months
  The investigators will use Likert scale for each question to evaluate the motivation to change. A score of 1 indicates that the participant has no intention to quit smoking and the score of 5 indicates that the participant is highly motivated. Evaluate the initial stage of change of the participant as judged by "Screening Questionnaire, Stage of Change". There is only 1 question.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Rochford, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Univeristy of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No